CLINICAL TRIAL: NCT05254106
Title: The Drug Eluting Devices French Safety Survey
Brief Title: The DETECT Project
Acronym: DETECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Collaborators: French-Speaking Vascular and Endovascular Surgery Society Support (Unknown); Boston Scientific Corporation (Industry); Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: RC20_0067
Record Dates: First submitted 2022-02-08; First posted 2022-02-24 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Femoropopliteal Atheromatous Lesions
Keywords: Femoropopliteal atheromatous lesions; endovascular revascularization; paclitaxel drug-eluting devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Paclitaxel drug-eluting devices: Patients treated by at least one paclitaxel drug-eluting balloon or stent after an endovascular femoropopliteal artery revascularization between October 2011 and December 2019 in France.
  Interventions: Device: Lower limb artery revascularization with paclitaxel-eluting device
- Non-drug-eluting devices: Patients exclusively treated by a non-drug-eluting balloon or stent after an endovascular femoropopliteal artery revascularization between October 2011 and December 2019 in France.

INTERVENTIONS:
Device: Lower limb artery revascularization with paclitaxel-eluting device — Lower limb artery revascularization with paclitaxel-eluting stent and/or paclitaxel-coated balloon
  Groups: Paclitaxel drug-eluting devices

SUMMARY:
This study aims to assess the all-cause mortality at 2 years of patients treated by a paclitaxel drug-eluting devices or non-drug-eluting devices after an endovascular femoropopliteal artery revascularization based on the French National Healthcare Data System (SNDS).

DETAILED DESCRIPTION:
Endovascular intervention is considered as a first-line treatment for femoropopliteal atheromatous lesions. During the 2000s, the superiority of auto-expandable stent compared to percutaneous transluminal angioplasty had been demonstrated, in terms of effectiveness. Over the past decade, paclitaxel drug-eluting balloons or stents were successfully assessed in order to prevent intimal hyperplasia and to treat restenosis.

Nevertheless, in 2018, Katsanos and al. reported in a meta-analysis a higher risk of death at 2 and 5 years for patients treated by a paclitaxel drug-eluting balloons or stents versus non-drug-eluting devices. This study presents many limitations despite being performed as a systematic review of randomized clinical trials. Since then, several studies have been conducted without any statistical trends in favor of a higher mortality in patients treated by drug-eluting stents or drug-coated balloons.

Analysis based on US or Germany databases in tens of thousands of patients has been published but individual data were unavailable. In France, there is no national report about the safety of paclitaxel drug-eluting devices prescribed in the case of endovascular femoropopliteal artery treatment. Therefore, this study aims to compare the risk of all-cause death of patients treated by paclitaxel-eluting devices versus non-drug-eluting devices in this indication at a national-scale using real-life data from SNDS.

This analysis of the SNDS database will allow (i) to identify all patients across France treated by endovascular intervention for a femoropopliteal revascularization and to know precisely the medical device used; (ii) to reduce confusion bias based on the characterization of patients thanks to their data of medical follow-up, treatment, hospitalization and LTD (long-term condition); (iii) to document their care pathway, especially drugs delivery and diagnosis associated to possible hospitalization, or to all-cause death, in order to compare the 1-, 2- and 5-years prognosis according to the medical device used.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old on day of hospital admission for the hereafter related surgical procedure
* Affiliated member to the French Social Security system
* Admitted in a French hospital, public or private, between October 2011 and December 2019
* Benefitting from an endovascular femoropopliteal surgical procedure coded with ≥ 1 of the 9 codes of the Common Classification of Medical Procedures (EEAF001, EEAF002, EEAF003, EEAF004, EEAF005, EEAF006, EEPF001, EEPF002, EELF002)
* Associated to the reimbursement by the health insurance scheme for one device of interest cited in the SAP (statistical analyses plan)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients included in this study were all patients identified in SNDS with an endovascular femoropopliteal artery intervention by non-drug-eluting balloon/stent or paclitaxel drug-eluting balloon/stent between October 2011 and December 2019 in France.
Sampling Method: Non-Probability Sample
Enrollment: 250000 (Estimated)
Dates: Start 2011-11-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Midterm mortality after the procedure of interest | 2 years
  All-cause death

SECONDARY OUTCOMES:
Short-term mortality after the procedure of interest | 1 year
  All-cause death
Long-term mortality after the procedure of interest | 5 years
  All-cause death
Adverse events after the procedure of interest | 1 year, 2 years, 5 years
  Hospitalization for coronary artery disease (myocardial infarction or coronary revascularization), cerebrovascular accident, transient ischemic attack, lower limb amputation (minor and major), a major adverse cardiovascular event (define as the composite of death, myocardial infarction, cerebrovascular accident, transient ischemic attack, major amputation), a major adverse limb event (define as the composite of a lower limb revascularization or a major amputation) or all-cause mortality.

CONTACTS AND LOCATIONS:
Locations (1):
- France, Whole Country, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wargny M, Leux C, Chatellier G, Coudol S, Gourraud PA, Goueffic Y. Mortality in a Nationwide Practice-Based Cohort Receiving Paclitaxel-Coated Devices for Lower Limb Peripheral Artery Disease. J Am Coll Cardiol. 2024 Apr 2;83(13):1207-1221. doi: 10.1016/j.jacc.2024.02.003. Epub 2024 Mar 25. PMID 38538200

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT05254106/SAP_000.pdf